CLINICAL TRIAL: NCT00998231
Title: Major Depression and Messenger RNAs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2009/15; 2009-A00405-52
Record Dates: First submitted 2009-07-29; First posted 2009-10-20 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Major Depressive Episode
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Major Depressive Episode (MDE) (Active Comparator): 20 subjects with major depressive episode will be included and followed during a 6 months interval which includes 4 visits (at the inclusion, 2 and 8 weeks later and finally 6 month later)
  Interventions: Biological: blood sample
- Control (Active Comparator): 20 subjects without major depressive episode will be included and followed during a 6 months interval which includes 4 visits (at the inclusion, 2 and 8 weeks later and finally 6 month later)
  Interventions: Biological: blood sample

INTERVENTIONS:
Biological: blood sample — Blood collections and peripheral blood mononuclear cells extraction will be operated after each evaluation and followed by RNA extraction, reverse transcription and gene expression quantification by real-time PCR.

SUMMARY:
Major Depressive Episode (MDE) affects nearly 15% of the general population. In a preliminary study, the investigators identified 12 genes whose expression was either altered between patient and control samples and/or between first patient samples and samples from the same patients obtained 8 weeks later. However, this study did not assess evolution of these alterations beyond an 8-week window and only 2 time points were considered. The investigators aim to compare gene expression difference for 21 candidate genes, of which 12 were already investigated, in 2 groups of subjects. MDE and control samples will be analyzed across a large time window to draw a better picture of the complex progression during MDE.

DETAILED DESCRIPTION:
Rational:

Major Depressive Episode (MDE) affects nearly 15% of the general population. To date, its pathophysiology remains unclear and treatment effects are often inconsistent. Therefore, it is challenging to make a valid prognosis for depression and identification of biomarkers is an important way of improving patient's treatment. Messenger RNAs (mRNAs) could be potential biological markers. Several studies have shown quantitative variations in peripheral blood mononuclear cells (PBMC) during MDE. These variations are state dependent and/or correlated with clinical measures.

In a preliminary study, the investigators identified 12 genes whose expression was either altered between patient and control samples and/or between first patient samples and samples from the same patients obtained 8 weeks later. However, this study did not assess evolution of these alterations beyond an 8 weeks window and only 2 time points were considered.

Objective:

the investigators aim to compare gene expression difference for 21 candidate genes, of which 12 were already investigated, in 2 groups of subjects. MDE and control samples will be analyzed across a large time window to draw a better picture of the complex progression during MDE.

Population and method:

This study is longitudinal and comparative. 20 subjects per group will be included and followed during a 6 months interval which includes 4 visits (at the inclusion, 2 and 8 weeks later and finally 6 month later). Clinical observations and psychometric scales will be used for evaluations. Blood collections and PBMCs extraction will be operated after each evaluation and followed by RNA extraction, reverse transcription and gene expression quantification by real-time PCR.

Expected results:

mRNA will be either over or under-expressed in patients during MDE in correlation with the clinical state. There will be no variation across time in control subjects. Comparison between MDE and control will show differences during MDE but not after clinical remission.

ELIGIBILITY:
Inclusion Criteria:

* Arm MDE:

  * Hamilton score on depression scale (HAMD-17) > 20;
  * No schizophrenia or bipolar disorder or disturbs delirious or evolutionary severe somatic pathology;
  * Taken care by a psychiatric department.
* Arm control:

  * No history of psychiatric pathology or evolutionary severe somatic pathology

Exclusion Criteria:

* Arm MDE:

  * Hamilton score on depression scale (HAMD-17) < or = 20;
  * With signs of schizophrenia or bipolar disorder or disturbs delirious;
  * With evolutionary severe somatic pathology.
* Arm control:

  * With signs of psychiatric pathology or evolutionary severe somatic pathology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-07; Primary Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
to compare gene expression difference for 21 candidate genes, of which 12 were already investigated, in 2 groups of subjects | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Raoul Belzeaux, Principal Investigator — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique-Hôpitaux de Marseille, Marseille, France